CLINICAL TRIAL: NCT01252472
Title: Diagnostic Imaging for Intraoperative Floppy Iris Syndrome
Brief Title: Flomax Study for Floppy Iris Syndrome
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roni Shtein, Assistant Professor of Ophthalmology and Visual Sciences, University of Michigan
Other Study IDs: HUM00039333
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Floppy Iris Syndrome
Keywords: Flomax; Floppy iris Syndrome; Tamsulosin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Flomax: Male patients scheduled for cataract surgery with current or past use of Flomax
- Control: Male adult patients scheduled for cataract surgery with no history of Flomax use

SUMMARY:
Some men who have a history of use of Tamsulosin (Flomax) are at risk for a condition called Intraoperative Floppy Iris Syndrome that can develop during otherwise routine cataract surgery. It is not fully understood why this condition develops or who is at risk for developing it. In this study the investigators will take pictures of the iris and iris blood vessels before cataract surgery. The investigators hope that the results of this study will provide a better understanding of how Intraoperative Floppy Iris Syndrome develops and give us a non-surgical way of figuring out who might develop this problem during surgery.

DETAILED DESCRIPTION:
Male patients scheduled for cataract surgery who are currently taking tamsulosin will be recruited into the study. Age-matched male control patients undergoing cataract surgery, without a history of using any a-adrenergic antagonist medication, will also be recruited. Careful diagnostic iris evaluation using iris Fluorescein Angiography (FA) and Anterior Segment Optical Coherence Tomography (AS-OCT) will be performed prior to cataract surgery. Intraoperative findings and surgical complications will be recorded in an effort to correlate preoperative diagnostic iris FA and AS-OCT findings with presence and severity of intraoperative floppy iris syndrome (IFIS). The investigators hypothesize that males on tamsulosin will have abnormal iris blood vessels on iris FA and altered iris morphology, consistent with iris atrophy, on AS-OCT that will correlate with presence of IFIS and help elucidate the pathophysiology of tamsulosin-induced IFIS.

Male patients scheduled for cataract surgery who are currently taking tamsulosin will be eligible for enrollment into the study if they have no other conditions that affect the iris vasculature and architecture (i.e. diabetes mellitus, glaucoma, pseudoexfoliation syndrome, history of prior eye surgery or eye trauma, use of eye drops other than artificial tears and normal preoperative drops). Control patients will be eligible if they have no history of use of any a-adrenergic antagonist (tamsulosin, alfuzosin, doxazosin, or terazosin). Patients who are interested in participating will be given a copy of the study consent form to take home with them. These patients will then be contacted by the study coordinator for further discussion of the study details. Study volunteers will be asked to come to the Kellogg Eye Center any time prior to their scheduled surgery. Volunteers will undergo the informed consent process, sign the consent form and be given a study identification number, linked to the patient in a de-identified fashion, that will be used exclusively for the study. The link of the study identification number and patient will be kept in a locked cabinet in the clinic coordinator's locked office. All patient study information will be collected and encoded according to HIPAA guidelines and institutional review board approval. The investigators plan to enroll 20 patients and 10 age-matched controls in a 12-month enrollment period.

* Iris Fluorescein Angiography (FA) will be performed in the surgical eye. The volunteer will be seated at the Heidelberg Spectralis (Heidelberg Engineering, Heidelberg, Germany) system. Sodium fluorescein dye (2mL of 25% solution) will be injected intravenously, and video images of the iris vasculature will be recorded as the fluorescent dye circulates through the iris blood vessels. The images will be digitally recorded and assigned the volunteer's study identification number. Data collected from this procedure includes circumferential extent of vascular filling (number of clock hours), radial extent of vascular filling (percent of iris radius), delay in iris circulation (time from dye injection to maximal filling of iris vasculature), blood vessel tortuosity and alterations in caliber. This procedure takes approximately 20 minutes.
* Anterior Segment Optical Coherence Tomography (AS-OCT) will be performed in the surgical eye. The volunteer will be seated at the Visante OCT (Carl Zeiss Meditec, Dublin, CA) in a room with standardized lighting. They will be instructed to look at a visual target within the instrument, and three high-resolution images of the anterior segment of the eye will be acquired and saved, identified only with the volunteer's study identification number. Data collected from this procedure includes iris leaflet thickness and pupil diameter in a controlled lighting situation. This procedure takes approximately 10 minutes.

Surgery will be performed according to the individual surgeon's preferences, including the use of any iris manipulation techniques that are clinically necessary. Surgical parameters will be recorded on a study visit form with the volunteer's study identification number:

* Pupil diameter will be measured with calipers at the beginning of surgery prior to incision, and at the end, after intraocular lens implantation, but prior to instillation of any miotic agents. These time points are before and after any intra-operative iris expansion techniques could be performed. The surgeon will also record whether he/she uses any iris expansion technique (i.e. iris hooks, Malyugin ring, non-standard pupil dilation medications), which one, and at what point in the procedure the technique was employed.
* Iris billowing will be graded as present or absent.
* Iris prolapse will be graded as present or absent.
* Surgical time from incision to dressing will be recorded.
* Surgical complications or any other surgical findings of interest to the surgeon will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years or older
* Scheduled for Cataract Surgery
* Current or Past use of Tamsulosin (flomax)
* Blue colored iris

For controls, no history of Flomax

Exclusion Criteria:

* Females
* Diabetes
* Glaucoma
* Use of medicated eye drops
* Trauma or prior surgery to the eye
* Black or brown iris

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male patients seen and scheduled for cataract surgery at the Kellogg eye Centers in Ann Arbor, Livonia and Brighton campuses.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative Floppy Iris Syndrome | during cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shtein, MD, Principal Investigator — University of Michigan Kellogg Eye Center
Locations (1):
- Kellogg Eye Center, 1000 Wall Street, Ann Arbor, Michigan, United States